CLINICAL TRIAL: NCT02036320
Title: A Non-dispensing Fit Evaluation of Investigational Limbal Ring Soft Contact Lenses With Polyvinylpyrrolidone (PVP) in Asian Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-5477
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-09

CONDITIONS: Vision Correction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A with additive printed limbal ring (Experimental): Each subject will insert the trial lens while being observed by a technician prior to assessment by the study investigator.
  Interventions: Device: etafilcon A
- etafilcon A (Active Comparator): Each subject will insert the trial lens while being observed by a technician prior to assessment by the study investigator.
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: etafilcon A — Each study subject will be exposed to both test lenses following a washout period of five minutes between test periods.

SUMMARY:
The purpose of this clinical trial is to compare the overall lens fit acceptance of two different soft contact lenses in an Asian population.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the statement of informed consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in the clinical protocol.
3. The subject must be an Asian female (self-reported).
4. The subject must be at least 18 years old and less than 41 years old.
5. The subject must meet two of the four East Asian anatomical categories (Appendix D) and have a prominent epicanthic fold to be classified East Asian ethnicity. For the purpose of this protocol, East Asian ethnicities may include: China, Japan, Korea, Taiwan, Vietnam, Hong Kong, Malaysia, and Singapore but are not inclusive of these regions.
6. The subject must be a habitual soft contact lens wearer. Habitual is defined as: at least one month of daily wear where the lenses are worn a minimum of six (6) hours per day and a minimum of three (3) days per week prior to enrollment in the study.
7. The subject's optimal non-vertexed spherical equivalent distance correction (based on their optimal sphero-cylinder refraction) must be between +2.00 D and -12.00 D.
8. Any cylinder power must be less than or equal to -1.00 D confirmed by refraction.
9. The subject must possess a functional/usable pair of spectacles and wear them to the visit (only if applicable-to the investigator's discretion).
10. The subject's best correctable visual acuity is 20/40 or better (OD and OS) at the baseline visit.

Exclusion Criteria:

1. Ocular or systemic allergies which might interfere with contact lens wear.
2. Ocular or systemic disease which might interfere with contact lens wear.
3. Any known hypersensitivity or allergic reaction to contact lenses or contact lens solutions.
4. Use of any ocular or topical medication.
5. Use of any systemic (oral) medication that is taken for an ocular condition which might interfere with contact lens wear.
6. Use of any systemic (oral) medication that is taken for a systemic condition which might interfere with the contact lens wear (this determination will be at the discretion of the investigator).
7. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities, bulbar injection or any other abnormalities of the cornea and/or conjunctiva which would contraindicate contact lens wear.
8. Rigid gas permeable or hybrid design (rigid gas permeable center and a soft lens skirt) contact lens wear within the past 30 days.
9. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
10. Any previous or planned (during duration of the study), ocular or intraocular surgery (e.g. radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), peripheral iridotomy, etc.)
11. Pregnancy or lactation.
12. Diabetes.
13. Infectious disease.
14. Habitual contact lens type is multifocal, monovision or worn as extended wear.
15. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
16. Suspicion of or recent history od alcohol or substance abuse.
17. History of serious mental illness.
18. History of seizures.
19. Employee or family member of the investigational clinic (e.g. Investigator, Coordinator, Technician).

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Berkeley, California
  - Fullerton, California
  - New York, New York
  - Cleveland, Ohio
  - Dallas, Texas
  - Houston, Texas
- Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 206 subjects were enrolled in this study. 16 subjects did not meet the eligibility criteria. 190 subjects were dispensed lenses and, 177 subjects completed all study visits without a major protocol deviation. 13 subjects were recorded as having protocol violations. No subjects were discontinued during this study.
Groups:
- Test 1/Test 2: Subjects who received test lens 1 first and then received test lens 2.
- Test 2/Test 1: Subjects who received test lens 2 first and then received test lens 1.
Period: Period 1
Arm/Group | Test 1/Test 2 | Test 2/Test 1
Started | 95 | 95
Completed | 95 | 95
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test 1/Test 2 | Test 2/Test 1
Started | 95 | 95
Completed | 95 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All subjects that were dispensed a test article during the study.
Arm/Group | Overall
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.75 (4.416)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 190
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 161
  Canada | 29

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Lens Fit Acceptance
Description: The number of subject eyes that were classified as having acceptable mechanical lens fit, with a slit lamp.
Time Frame: 15 mins post insertion
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Test 1: Subjects that received Test lens 1 during the first or second period of the study.
- Test 2: Subjects that received Test lens 2 during the first or second period of the study.
Arm/Group | Test 1 | Test 2
Number analyzed (Participants) | 177 | 177
Number analyzed (Eyes) | 354 | 354
Eyes | 345 | 337

2. Primary Outcome: Cosmetic Lens Fit Acceptance
Description: The number of subject eyes that were classified as having acceptable cosmetic lens fit in primary gaze, without a slit lamp.
Time Frame: 15 mins post insertion
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Test 1 | Test 2
Number analyzed (Participants) | 177 | 177
Number analyzed (Eyes) | 354 | 354
Eyes | 349 | 349

3. Primary Outcome: Lens Does Not Exhibit "Hula Hoop" Effect
Description: The number of subjects that did not exhibit a "hula hoop" effect as recorded by Eye Care Practitioner (ECP) judgment of acceptable physiology, in primary gaze, without a slit lamp.
Time Frame: 15 mins post insertion
Population: The analysis population consists of subjects that completed all study visits, without a major protocol deviation
Measure: Number; unit: Subject
Arm/Group | Test 1 | Test 2
Number analyzed (Participants) | 177 | 177
Subject | 176 | 176

ADVERSE EVENTS:
Arm/Group | Test 1 | Test 2
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/95
Other Adverse Events (participants affected / at risk) | 0/95 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days